CLINICAL TRIAL: NCT05724836
Title: Prospective Carotid Artery Stenosis Trial
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Young M. Erben, Principal Investigator, Mayo Clinic
Other Study IDs: 23-000525
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Patients With Any Degree of Carotid Artery Stenosis and Vulnerable Features in the Carotid Artery Plaque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Researchers are collecting information and blood from subjects undergoing carotid artery interventions.

ELIGIBILITY:
Inclusion Criteria:

* All subjects undergoing carotid artery intervention that presents to our clinic

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing carotid artery intervention
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Biospecimen Acquisition | 1 month
  Number of biospecimens collected

CONTACTS AND LOCATIONS:
Overall Officials: Young M Erben, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials